CLINICAL TRIAL: NCT06837402
Title: Epidemiology of Non- Invasive Mechanical Ventilation in Argentina: a Multicenter Observational Study
Acronym: EpVAr-VMNI
Status: Enrolling by invitation | Type: Observational
Sponsor: Argentinian Intensive Care Society (Other)
Responsible Party: Principal Investigator, Gustavo Plotnikow, Respiratory Therapist, Argentinian Intensive Care Society
Other Study IDs: 14770
Record Dates: First submitted 2025-02-11; First posted 2025-02-20 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Respiration, Artificial; Noninvasive Ventilation; Intensive Care Units
Keywords: mechanical ventilation; acute respiratory failure; noninvasive ventilation; intensive care unit
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction Non-invasive mechanical ventilation (NIMV) is a fundamental strategy in the management of acute respiratory failure, preventing intubation and reducing complications. However, the epidemiology of its use in Argentina is not well understood, motivating this study.

Justification Unequal access to ICU resources in Argentina affects the quality of care. This study aims to describe the implementation, effectiveness, and outcomes of NIMV across different regions of the country to improve clinical decision-making and healthcare policies.

Objectives

* Primary: Analyze the survival of ICU patients receiving NIMV.
* Secondary: Evaluate success/failure factors, regional disparities in resource availability, the impact of healthcare staff training, comparison between public and private sectors, and establish a national database.

Methods Study Design Observational, multicenter, prospective, and analytical study. Both public and private hospitals in Argentina will be included. Data will be collected over seven months, with patient follow-up until discharge or death.

Study Population Adult patients (>18 years) admitted to the ICU requiring NIMV for acute respiratory failure or as part of weaning from invasive mechanical ventilation.

Inclusion Criteria

* Age >18 years.
* Use of NIMV in the ICU for respiratory failure or during weaning.
* Signed informed consent.

Exclusion Criteria

* Patients using home NIMV without exacerbation.
* Patients without acute respiratory impairment.

Data Collection and Management

* Data will be recorded using an electronic form in RedCap®, with restricted access.
* Confidentiality will be ensured through alphanumeric coding.
* A monitoring committee will supervise data quality.

Statistical Analysis

* Continuous variables: Mean and standard deviation or median and interquartile range.
* Comparisons: Student's t-test, Mann-Whitney U test, Chi² test, or Fisher's exact test.
* Multivariate models: Logistic regression and Kaplan-Meier survival analysis.

Bias Control and Data Quality Strategies will be implemented to minimize selection, information, and investigator bias. Data will be periodically reviewed by the monitoring committee.

Study Feasibility The study is supported by the British Hospital of Buenos Aires and the Argentine Society of Intensive Care Medicine, ensuring its viability.

Ethical Considerations The study will comply with national and international health research regulations, ensuring participant confidentiality.

Publication and Funding The study will be funded by the Argentine Society of Intensive Care Medicine, with no external financial support. Authorship in publications will depend on the number of patients included per center.

Conclusion This study aims to generate key information on NIMV use in Argentina, optimizing its application and improving ICU care nationwide.

DETAILED DESCRIPTION:
Background and Rationale Non-invasive mechanical ventilation (NIMV) has become a crucial treatment in managing acute respiratory failure, preventing the need for endotracheal intubation and its associated complications. Numerous studies have demonstrated that timely and appropriate NIMV use reduces mortality, decreases the incidence of ventilator-associated pneumonia, and minimizes hospital length of stay. However, the epidemiology of NIMV use in Argentina remains largely undocumented, particularly regarding regional disparities in access, implementation, and patient outcomes.

This multicenter observational study aims to fill this knowledge gap by analyzing NIMV utilization in intensive care units (ICUs) across Argentina. The study will evaluate patient characteristics, clinical outcomes, and factors influencing NIMV success or failure. Additionally, it will assess the impact of healthcare staff training and the differences between public and private healthcare settings.

Study Objectives Primary Objective

- Analyze the survival rates of ICU patients receiving NIMV.

Secondary Objectives

* Identify factors associated with NIMV success or failure, including the need for intubation.
* Describe demographic and clinical characteristics of patients requiring NIMV.
* Compare mortality rates between successful and failed NIMV cases.
* Evaluate regional disparities in resource availability and NIMV usage.
* Analyze the impact of staff training levels on patient outcomes.
* Compare NIMV practices between public and private hospitals.
* Establish a national database to facilitate ongoing assessment of NIMV in Argentina.

Study Design This is a prospective, multicenter, observational, and analytical study that will collect data from ICUs in both public and private hospitals across different regions of Argentina. The study will be conducted over seven months to capture seasonal variations in respiratory diseases. All enrolled patients will be followed until discharge or death.

Population and Setting The study will include adult patients (≥18 years old) admitted to ICUs and requiring NIMV for acute respiratory failure or as part of weaning from invasive mechanical ventilation (IMV). Participating hospitals must have the capacity to provide NIMV and record detailed patient data.

Eligibility Criteria

Inclusion Criteria:

* Patients ≥18 years old requiring NIMV in ICU for acute respiratory failure (hypoxemic, hypercapnic, or mixed) or as part of IMV weaning.
* Patients receiving palliative NIMV or as part of end-of-life care.
* Patients requiring increased duration or level of NIMV support due to worsening condition.
* Signed informed consent from the patient or a legal representative.

Exclusion Criteria:

* Patients using home NIMV for chronic respiratory conditions (e.g., COPD, neuromuscular diseases, obesity hypoventilation syndrome) without acute respiratory deterioration.
* Patients without acute respiratory distress at ICU admission.

Data Collection and Variables Data Management System

* Data will be collected using an electronic form in RedCap® with restricted access.
* Each participating ICU will have a designated site coordinator responsible for data collection and entry.
* To ensure data accuracy, a monitoring committee will review a random 5% sample of enrolled patients.

Key Variables Baseline Data

* Demographics: Age, sex, weight, height.
* ICU admission data: Date of hospital and ICU admission.
* Charlson Comorbidity Index and APACHE II score at ICU admission.
* Previous NIMV or oxygen therapy use (home or pre-ICU).

NIMV Implementation

* Date of NIMV initiation in ICU.
* Initial arterial blood gas (ABG) values: pH, PaCO₂, PaO₂, SaO₂, FiO₂.
* Primary reason for NIMV: COPD exacerbation, asthma, pneumonia, ARDS, post-operative respiratory failure, cardiogenic pulmonary edema, neuromuscular disease, etc.
* Ventilator settings: Mode (e.g., PSV, PCV), inspiratory pressure, PEEP, FiO₂, respiratory rate, tidal volume.
* Interface used: Helmet, oronasal mask, nasal mask, mouthpiece.
* Humidification use (active/passive).
* Adjunct therapies: Sedation, analgesia, high-flow nasal oxygen (HFNO).

Monitoring and Outcomes

* Daily ABG values and ventilator settings during NIMV use.
* Signs of respiratory distress: Tachypnea, accessory muscle use, paradoxical breathing.
* Complications: Facial pressure ulcers, barotrauma, pneumonia, gastric distension.
* Failure criteria: Need for intubation or death during NIMV.
* Length of NIMV use and ICU/hospital stay duration.
* Mortality at day 28 and at hospital discharge.
* Final disposition: Discharge to home, rehabilitation center, or another hospital unit.

Statistical Analysis

* Descriptive statistics:
* Continuous variables: Mean ± SD or median (IQR).
* Categorical variables: Frequency and percentages.
* Comparative analysis:
* Student's t-test or Mann-Whitney U test for continuous variables.
* Chi-square test or Fisher's exact test for categorical variables.
* Multivariate analysis:
* Logistic regression to identify predictors of NIMV failure.
* Kaplan-Meier survival analysis and Cox proportional hazards model to assess survival outcomes.
* Missing data handling: Patients with >10% missing key variables will be excluded from the final analysis.
* Software: All statistical analyses will be performed using R 4.3.3, with ggplot2 for visualizations and Survival package for survival analysis.

Bias Control and Quality Assurance

* Selection bias: Consecutive patient recruitment to minimize inclusion bias.
* Information bias: Standardized electronic data collection with training for investigators.
* Investigator bias: Use of predefined diagnostic criteria and cut-off values.

Ethical Considerations

* The study will comply with international research ethics standards (Helsinki Declaration, ICH-GCP).
* Data will be anonymized and securely stored, following Argentina's Data Protection Law (25.326/00).
* Ethical approval will be obtained from the Ethics Committee of the British Hospital of Buenos Aires and participating institutions.

Study Feasibility

* The study will be coordinated by the British Hospital of Buenos Aires with support from the Argentine Society of Intensive Care Medicine (SATI).
* No external funding; the study is supported by SATI.
* Participating centers will be invited via SATI networks and social media, with a structured training program to ensure compliance with data collection protocols.

Conclusion This study will provide essential insights into NIMV epidemiology in Argentina, helping to optimize its implementation and improve ICU care nationwide. By identifying key predictors of success or failure, the study will contribute to evidence-based clinical practice and inform national health policies regarding ventilatory support strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Requirement of NIMV in ICU due to acute respiratory failure (hypoxemic or hypercapnic or mixed) or as part of the process of weaning from mechanical ventilation.
* Patients who receive NIMV as a palliative or as part of end-of-life care.
* Patients as a routine treatment who require an increase in the time of use, or the level of support, or both due to increased demand.
* Informed consent signed by the patient or his/her legal representative in the event that the patient is incapacitated.

Exclusion Criteria:

* Patients admitted to the ICU with NIV as standard treatment for chronic lung disease, neuromuscular disease, obstructive sleep apnea-hypopnea syndrome, or obesity hypoventilation syndrome without additional respiratory compromise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU with NIMV requirements
Sampling Method: Non-Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
ICU Mortality | 28 days
  Death that occurs during Hospital stay
Hospital Mortality | 28 days
  Death that occurs during ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Plotnikow, RT, Principal Investigator — Hospital Británico
Locations (1):
- Hospital Británico de Buenos Aires, CABA, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rochwerg B, Brochard L, Elliott MW, Hess D, Hill NS, Nava S, Navalesi P Members Of The Steering Committee, Antonelli M, Brozek J, Conti G, Ferrer M, Guntupalli K, Jaber S, Keenan S, Mancebo J, Mehta S, Raoof S Members Of The Task Force. Official ERS/ATS clinical practice guidelines: noninvasive ventilation for acute respiratory failure. Eur Respir J. 2017 Aug 31;50(2):1602426. doi: 10.1183/13993003.02426-2016. Print 2017 Aug. PMID 28860265
- [Background] Chawla R, Dixit SB, Zirpe KG, Chaudhry D, Khilnani GC, Mehta Y, Khatib KI, Jagiasi BG, Chanchalani G, Mishra RC, Samavedam S, Govil D, Gupta S, Prayag S, Ramasubban S, Dobariya J, Marwah V, Sehgal I, Jog SA, Kulkarni AP. ISCCM Guidelines for the Use of Non-invasive Ventilation in Acute Respiratory Failure in Adult ICUs. Indian J Crit Care Med. 2020 Jan;24(Suppl 1):S61-S81. doi: 10.5005/jp-journals-10071-G23186. PMID 32205957
- [Background] Fujishima S. Guideline-based management of acute respiratory failure and acute respiratory distress syndrome. J Intensive Care. 2023 Mar 10;11(1):10. doi: 10.1186/s40560-023-00658-3. PMID 36895001
- [Background] Nava S, Navalesi P, Conti G. Time of non-invasive ventilation. Intensive Care Med. 2006 Mar;32(3):361-70. doi: 10.1007/s00134-005-0050-0. Epub 2006 Feb 14. PMID 16477416
- [Background] Klefti G, Hill AT. The benefits of non-invasive ventilation for Community-Acquired Pneumonia: A meta-analysis. QJM. 2020 Mar 30:hcaa106. doi: 10.1093/qjmed/hcaa106. Online ahead of print. PMID 32227219
- [Background] Burns KEA, Stevenson J, Laird M, Adhikari NKJ, Li Y, Lu C, He X, Wang W, Liang Z, Chen L, Zhang H, Friedrich JO. Non-invasive ventilation versus invasive weaning in critically ill adults: a systematic review and meta-analysis. Thorax. 2022 Aug;77(8):752-761. doi: 10.1136/thoraxjnl-2021-216993. Epub 2021 Oct 29. PMID 34716282
- [Background] Osadnik CR, Tee VS, Carson-Chahhoud KV, Picot J, Wedzicha JA, Smith BJ. Non-invasive ventilation for the management of acute hypercapnic respiratory failure due to exacerbation of chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2017 Jul 13;7(7):CD004104. doi: 10.1002/14651858.CD004104.pub4. PMID 28702957
- [Background] Farhan H, Moreno-Duarte I, Latronico N, Zafonte R, Eikermann M. Acquired Muscle Weakness in the Surgical Intensive Care Unit: Nosology, Epidemiology, Diagnosis, and Prevention. Anesthesiology. 2016 Jan;124(1):207-34. doi: 10.1097/ALN.0000000000000874. PMID 26445385
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Dowdy DW, Eid MP, Sedrakyan A, Mendez-Tellez PA, Pronovost PJ, Herridge MS, Needham DM. Quality of life in adult survivors of critical illness: a systematic review of the literature. Intensive Care Med. 2005 May;31(5):611-20. doi: 10.1007/s00134-005-2592-6. Epub 2005 Apr 1. PMID 15803303
- [Background] Combes A, Costa MA, Trouillet JL, Baudot J, Mokhtari M, Gibert C, Chastre J. Morbidity, mortality, and quality-of-life outcomes of patients requiring >or=14 days of mechanical ventilation. Crit Care Med. 2003 May;31(5):1373-81. doi: 10.1097/01.CCM.0000065188.87029.C3. PMID 12771605
- [Background] Cuthbertson BH, Hull A, Strachan M, Scott J. Post-traumatic stress disorder after critical illness requiring general intensive care. Intensive Care Med. 2004 Mar;30(3):450-5. doi: 10.1007/s00134-003-2004-8. Epub 2003 Sep 5. PMID 12961065
- [Background] Jubran A, Lawm G, Duffner LA, Collins EG, Lanuza DM, Hoffman LA, Tobin MJ. Post-traumatic stress disorder after weaning from prolonged mechanical ventilation. Intensive Care Med. 2010 Dec;36(12):2030-7. doi: 10.1007/s00134-010-1972-8. Epub 2010 Jul 27. PMID 20661726
- [Background] Jubran A, Lawm G, Kelly J, Duffner LA, Gungor G, Collins EG, Lanuza DM, Hoffman LA, Tobin MJ. Depressive disorders during weaning from prolonged mechanical ventilation. Intensive Care Med. 2010 May;36(5):828-35. doi: 10.1007/s00134-010-1842-4. Epub 2010 Mar 16. PMID 20232042
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] MacIntyre NR, Cook DJ, Ely EW Jr, Epstein SK, Fink JB, Heffner JE, Hess D, Hubmayer RD, Scheinhorn DJ; American College of Chest Physicians; American Association for Respiratory Care; American College of Critical Care Medicine. Evidence-based guidelines for weaning and discontinuing ventilatory support: a collective task force facilitated by the American College of Chest Physicians; the American Association for Respiratory Care; and the American College of Critical Care Medicine. Chest. 2001 Dec;120(6 Suppl):375S-95S. doi: 10.1378/chest.120.6_suppl.375s. No abstract available. PMID 11742959
- [Background] Nava S, Ambrosino N, Rubini F, Fracchia C, Rampulla C, Torri G, Calderini E. Effect of nasal pressure support ventilation and external PEEP on diaphragmatic activity in patients with severe stable COPD. Chest. 1993 Jan;103(1):143-50. doi: 10.1378/chest.103.1.143. PMID 8417869
- [Background] Appendini L, Patessio A, Zanaboni S, Carone M, Gukov B, Donner CF, Rossi A. Physiologic effects of positive end-expiratory pressure and mask pressure support during exacerbations of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1994 May;149(5):1069-76. doi: 10.1164/ajrccm.149.5.8173743.
- [Background] Mehta S, Hill NS. Noninvasive ventilation. Am J Respir Crit Care Med. 2001 Feb;163(2):540-77. doi: 10.1164/ajrccm.163.2.9906116. No abstract available. PMID 11179136
- [Background] Rathgeber J, Schorn B, Falk V, Kazmaier S, Spiegel T, Burchardi H. The influence of controlled mandatory ventilation (CMV), intermittent mandatory ventilation (IMV) and biphasic intermittent positive airway pressure (BIPAP) on duration of intubation and consumption of analgesics and sedatives. A prospective analysis in 596 patients following adult cardiac surgery. Eur J Anaesthesiol. 1997 Nov;14(6):576-82. doi: 10.1046/j.1365-2346.1994.00178.x. PMID 9466092
- [Background] Criner GJ, Tzouanakis A, Kreimer DT. Overview of improving tolerance of long-term mechanical ventilation. Crit Care Clin. 1994 Oct;10(4):845-66. PMID 8000930
- [Background] Esteban A, Anzueto A, Frutos F, Alia I, Brochard L, Stewart TE, Benito S, Epstein SK, Apezteguia C, Nightingale P, Arroliga AC, Tobin MJ; Mechanical Ventilation International Study Group. Characteristics and outcomes in adult patients receiving mechanical ventilation: a 28-day international study. JAMA. 2002 Jan 16;287(3):345-55. doi: 10.1001/jama.287.3.345. PMID 11790214
- [Background] Esteban A, Ferguson ND, Meade MO, Frutos-Vivar F, Apezteguia C, Brochard L, Raymondos K, Nin N, Hurtado J, Tomicic V, Gonzalez M, Elizalde J, Nightingale P, Abroug F, Pelosi P, Arabi Y, Moreno R, Jibaja M, D'Empaire G, Sandi F, Matamis D, Montanez AM, Anzueto A; VENTILA Group. Evolution of mechanical ventilation in response to clinical research. Am J Respir Crit Care Med. 2008 Jan 15;177(2):170-7. doi: 10.1164/rccm.200706-893OC. Epub 2007 Oct 25. PMID 17962636
- [Background] Esteban A, Frutos-Vivar F, Muriel A, Ferguson ND, Penuelas O, Abraira V, Raymondos K, Rios F, Nin N, Apezteguia C, Violi DA, Thille AW, Brochard L, Gonzalez M, Villagomez AJ, Hurtado J, Davies AR, Du B, Maggiore SM, Pelosi P, Soto L, Tomicic V, D'Empaire G, Matamis D, Abroug F, Moreno RP, Soares MA, Arabi Y, Sandi F, Jibaja M, Amin P, Koh Y, Kuiper MA, Bulow HH, Zeggwagh AA, Anzueto A. Evolution of mortality over time in patients receiving mechanical ventilation. Am J Respir Crit Care Med. 2013 Jul 15;188(2):220-30. doi: 10.1164/rccm.201212-2169OC. PMID 23631814
- [Background] Estenssoro E, Plotnikow G, Loudet CI, Rios FG, Kanoore Edul VS, Andrian M, Romero I, Sagardia J, Bezzi M, Mandich V, Groer C, Torres S, Orlandi C, Rubatto Birri PN, Valenti MF, Cunto E, Saenz MG, Tiribelli N, Aphalo V, Betttini L, Reina R, Dubin A; Grupo de investigadores del estudio SATICOVID-19. [Structural capacity, technological human resources and mechanical ventilation requirements in 58 intensive care units in Argentina during the SARS-CoV-2 pandemic. A SATICOVID-19 Study]. Medicina (B Aires). 2022;82(1):35-46. Spanish. PMID 35037859
- [Background] Plotnikow GA, Gogniat E, Accoce M, Navarro E, Dorado JH; EpVAr study group. Epidemiology of mechanical ventilation in Argentina. The EpVAr multicenter observational study. Med Intensiva (Engl Ed). 2022 Jul;46(7):372-382. doi: 10.1016/j.medine.2022.05.002. Epub 2022 May 31. PMID 35660286
- [Background] Dorado JH, Navarro E, Plotnikow GA, Gogniat E, Accoce M; EpVAr Study Group. Epidemiology of Weaning From Invasive Mechanical Ventilation in Subjects With COVID-19. Respir Care. 2023 Jan;68(1):101-109. doi: 10.4187/respcare.09925. Epub 2022 Nov 15. PMID 36379638
- [Background] R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. R Core Team (2017). [cited 21 Dec 2024]. URL: https://www.r-project.org/
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Charlson ME, Charlson RE, Peterson JC, Marinopoulos SS, Briggs WM, Hollenberg JP. The Charlson comorbidity index is adapted to predict costs of chronic disease in primary care patients. J Clin Epidemiol. 2008 Dec;61(12):1234-1240. doi: 10.1016/j.jclinepi.2008.01.006. Epub 2008 Jul 10. PMID 18619805
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Metlay JP, Waterer GW, Long AC, Anzueto A, Brozek J, Crothers K, Cooley LA, Dean NC, Fine MJ, Flanders SA, Griffin MR, Metersky ML, Musher DM, Restrepo MI, Whitney CG. Diagnosis and Treatment of Adults with Community-acquired Pneumonia. An Official Clinical Practice Guideline of the American Thoracic Society and Infectious Diseases Society of America. Am J Respir Crit Care Med. 2019 Oct 1;200(7):e45-e67. doi: 10.1164/rccm.201908-1581ST. PMID 31573350
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Estenssoro E, Gonzalez I, Plotnikow GA. Post-pandemic acute respiratory distress syndrome: A New Global Definition with extension to lower-resource regions. Med Intensiva (Engl Ed). 2024 May;48(5):272-281. doi: 10.1016/j.medine.2024.01.011. Epub 2024 Apr 20. PMID 38644108
- [Background] Toro AC, Escobar LM, Franco JG, Diaz-Gomez JL, Munoz JF, Molina F, Bejarano J, Yepes D, Navarro E, Garcia A, Ely WE, Esteban A. [Spanish version of the CAM-ICU (Confusion Assessment Method for the Intensive Care Unit). Pilot study of validation]. Med Intensiva. 2010 Jan-Feb;34(1):14-21. doi: 10.1016/j.medin.2009.07.002. Epub 2009 Sep 30. Spanish. PMID 20233574
- [Background] Vicente-Herrero MT, Delgado-Bueno S, Bandrés-Moyá F, Ramírez-Iñiguez-de- la-Torre MV, Capdevilla-García L. Valoración del dolor. Revisión comparativa de escalas y cuestionarios. Revista de la Sociedad Española del Dolor 2018; 25(4): 228-236.
- [Background] Teasdale G, Jennett B. Assessment of coma and impaired consciousness. A practical scale. Lancet. 1974 Jul 13;2(7872):81-4. doi: 10.1016/s0140-6736(74)91639-0. No abstract available. PMID 4136544